CLINICAL TRIAL: NCT05452798
Title: A Retrospective Non-interventional Study of Breast Cancer Patients Diagnosed With HR+/HER2- Locally Advanced or Metastatic Breast Cancer Treated With Palbociclib in Denmark
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481176
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: Metastatic Breast Cancer; HR+/ HER2-
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The objective is to retrospectively describe and assess clinical and demographical characteristics, treatment patterns in a real-world (RW) setting of patients with HR+/HER2- (hormone receptor positive/human epidermal growth factor receptor 2 negative) locally advanced or metastatic breast cancer receiving palbociclib in combination treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer (International Statistical Classification of Diseases and Related Health Problems, 10th Revision [ICD-10]: ICD-10 code for patients with breast cancer [DC50])
* A diagnosis of HR+/HER2- locally advanced or metastatic breast cancer
* Initiated treatment with palbociclib as either 1st or 2nd line treatment between 01 January 2017 and 31 December 2020
* Inclusion date: Date of relapse/stage IV disease/progression leading to initiation of palbociclib+AI/progression leading to initiation of palbociclib+fulvestrant

Exclusion Criteria:

* There are no exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HR+/HER2- locally advanced or metastatic breast cancer treated with palbociclib (1st or 2nd line between 01 Jan 2017- 31 Dec 2020).
Sampling Method: Non-Probability Sample
Enrollment: 1054 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Danish Breast Cancer Group, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with hormone receptor positive/human epidermal growth factor receptor 2 negative (HR+/HER2-) locally advanced or metastatic breast cancer (BC) who initiated treatment with palbociclib in Denmark as either first or second line treatment between 01 January 2017 and 31 December 2020 were observed. Data was collected retrospectively from Danish Breast Cancer Group (DBCG) registry. Data analysis was performed over approximately 5 months in this study.
Groups:
- Palbociclib: Participants with HR+/HER2- locally advanced or metastatic BC who initiated treatment with palbociclib as first or second line treatment between 01 January 2017 and 31 December 2020 were observed in this retrospective study.
Period: Overall Study
Arm/Group | Palbociclib
Started | 1054
Completed | 1054
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all eligible participants with HR+/HER2- locally advanced or metastatic BC who initiated treatment with palbociclib as first or second line treatment between 01 January 2017 and 31 December 2020.
Arm/Group | Palbociclib
Number analyzed (Participants) | 1054
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 66.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 1054
  Sex: Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) for Participants Who Received Palbociclib in Combination With Aromatase Inhibitor (AI)
Description: PFS was defined as the time from the index date to progression or death, whichever occurred first. Progression of disease was based on scans and blood testing results. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). Index date was date of relapse or stage IV disease. Stage IV disease means that the cancer has spread to distant parts of the body. Kaplan-Meier method was used for analysis.
Time Frame: From index date until the first documentation of disease progression or death or censoring date of 07-Mar-2022 (maximum up to 5.2 years)
Population: Analysis was performed on participants with HR+/HER2- locally advanced or metastatic BC who initiated treatment with palbociclib in combination with AI between 01 January 2017 and 31 December 2020.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 525
Months | 27.4 [12.4 to 57.3]

2. Secondary Outcome: Overall Survival (OS) in Participants Who Received Palbociclib in Combination With AI
Description: OS was defined as the date of metastatic breast cancer diagnosis until death of any cause. Participants were censored for OS by 01-May-2022. Stage IV disease means that the cancer has spread to distant parts of the body.
Time Frame: From date of metastatic breast cancer diagnosis until death due to any cause or censoring date of 01-May-2022 (approximately 6 years)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 525
Months | 54.2 [29.5 to 72.3]

3. Secondary Outcome: Progression-Free Survival (PFS) for Participants Who Received Palbociclib in Combination With Fulvestrant
Description: PFS was defined as the time from the index date to progression or death, whichever occurred first. Progression of disease was based on scans and blood testing results. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Index date was date of relapse or stage IV disease. Stage IV disease means that the cancer has spread to distant parts of the body.
Time Frame: as for outcome 1
Population: Analysis was performed on participants with HR+/HER2- locally advanced or metastatic BC who initiated treatment with palbociclib in combination with fulvestrant between 01 January 2017 and 31 December 2020.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 524
Months | 14.9 [5.9 to 30.3]

4. Secondary Outcome: Time on Treatment (ToT) for Participants Who Received Palbociclib in Combination With Fulvestrant
Description: ToT is defined as date of palbociclib treatment start to date of treatment stop with palbociclib.
Time Frame: From start date of study treatment until stop date of treatment (maximum up to 5.2 years)
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 524
Months | 11.2 [3.7 to 23.7]

5. Primary Outcome: Time on Treatment (ToT) for Participants Who Received Palbociclib in Combination With Aromatase Inhibitor (AI)
Description: ToT was defined as date of palbociclib treatment start to date of treatment stop with palbociclib.
Time Frame: From start date of palbociclib treatment until stop date of palbociclib treatment (maximum up to 5.2 years)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 525
Months | 18.5 [7 to 41.1]

6. Secondary Outcome: OS in Participants Who Received Palbociclib in Combination With Fulvestrant
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Palbociclib
Number analyzed (Participants) | 524
Months | 32.9 [19.0 to 56.0]

7. Secondary Outcome: Number of Participants According to First Subsequent Post-Palbociclib Treatment Upon Progression
Description: Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Number of participants as per first subsequent post-palbociclib therapy upon disease progression was described in this outcome measure.
Time Frame: At progression (anytime between 01 January 2017 and 31 December 2020 [maximum up to 4 years])
Population: Analysis was performed on participants with HR+/HER2- locally advanced or metastatic BC who initiated treatment with palbociclib in combination with AI or fulvestrant between 01 January 2017 and 31 December 2020. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 667
Participants
  Chemotherapy | 350
  Endocrine therapy | 315
  Other treatment | 2

8. Secondary Outcome: Number of Participants According to Type of Metastases
Description: Number of participants according to type of metastases (visceral, non-visceral, both visceral and non-visceral and inoperable locally-advanced breast cancer [ILABC]) is presented in this outcome measure.
Time Frame: At Baseline (anytime between 01 January 2017 and 31 December 2020 [maximum up to 4 years])
Population: Analysis was performed on participants with HR+/HER2- locally advanced or metastatic BC who initiated treatment with palbociclib as first or second line treatment between 01 January 2017 and 31 December 2020.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 1054
Participants
  Visceral metastases | 105
  Non-visceral metastases | 405
  Both visceral and non-visceral metastases | 530
  Inoperable locally advanced breast cancer (ILABC) | 14

9. Secondary Outcome: Number of Participants According to Number of Metastases
Description: Number of participants according to number of metastases (0,1,2,greater than [>] 2) is presented in this outcome measure.
Time Frame: At Baseline (anytime between 01 January 2017 and 31 December 2020 [maximum up to 4 years])
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 1054
Participants
  0 | 14
  1 | 375
  2 | 303
  > 2 | 362

10. Secondary Outcome: Number of Participants According to Location of Metastases
Description: Number of participants according to location of metastases (skin, bone, lung, liver, central nervous system [CNS], other) is presented in this outcome measure. One participant may have more than one location of metastases.
Time Frame: At Baseline (anytime between 01 January 2017 and 31 December 2020 [maximum up to 4 years])
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 1054
Participants
  Skin | 80
  Bone | 790
  Lung | 417
  Liver | 268
  Central nervous system (CNS) | 41
  Other | 480

11. Secondary Outcome: Number of Participants Who Underwent Surgery
Description: Number of participants who underwent surgery were described.
Time Frame: At Baseline (anytime between 01 January 2017 and 31 December 2020 [maximum up to 4 years])
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 1054
Participants | 96

12. Secondary Outcome: Number of Participants According to Type of Adjuvant Treatment
Description: Participants who received adjuvant treatment (endocrine therapy, taxane, cyclophosphamide and epirubicin, unknown and other) were described in this outcome measure. One participant may have received more than one type of adjuvant treatment.
Time Frame: At Baseline (anytime between 01 January 2017 and 31 December 2020 [maximum up to 4 years])
Population: Analysis was performed on participants with HR+/HER2- locally advanced or metastatic BC who initiated treatment with palbociclib as first or second line treatment between 01 January 2017 and 31 December 2020. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 784
Participants
  Endocrine therapy | 552
  Taxane | 202
  Cyclophosphamide and epirubicin | 194
  Unknown | 176
  Other | 122

13. Secondary Outcome: Number of Participants With De Novo and Recurrent Metastatic Breast Cancer
Description: Participants who had de novo and recurrent metastatic breast cancer were reported in this outcome measure.
Time Frame: At Baseline (anytime between 01 January 2017 and 31 December 2020 [maximum up to 4 years])
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib
Number analyzed (Participants) | 1054
Participants
  Recurrent metastatic breast cancer | 784
  De Novo metastatic breast cancer | 270

14. Secondary Outcome: Median Time From Initial Breast Cancer Diagnosis to Relapse
Description: Median time from initial breast cancer diagnosis (incidence date) to relapse is reported in this outcome measure.
Time Frame: At Baseline (anytime between 01 January 2017 and 31 December 2020 [maximum up to 4 years])
Population: as for outcome 8
Measure: Median (Full Range); unit: years
Arm/Group | Palbociclib
Number analyzed (Participants) | 1054
years | 5.2 [NA to NA] — Only median was planned as per statistical analysis plan.

ADVERSE EVENTS:
Time Frame: All-cause mortality: From date of metastatic breast cancer diagnosis until the end of follow-up (approximately 6 years). Data for non-serious adverse events and serious adverse events (SAEs) were not collected and evaluated during the study; hence timeframe is not applicable for non-SAEs and SAEs.
Description: This observational retrospective study retrieved data from DBCG registry. In these data sources, individual participant data were not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event could not be met, hence adverse events data were not collected and reported.
Arm/Group | Palbociclib
All-Cause Mortality (participants affected / at risk) | 525/1054
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT05452798/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT05452798/SAP_001.pdf